CLINICAL TRIAL: NCT02609282
Title: Pilot Study to Assess the Impact of Hourly Prompts, Delivered by Microsoft Outlook, on Reducing Prolonged Sitting at Work
Brief Title: The Impact of Hourly Prompts on Reducing Prolonged Sitting at Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: Scottish Centre for Healthy Working Lives (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GlasgowCU
Record Dates: First submitted 2015-09-10; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Sedentary Lifestyle
Keywords: Sedentary behaviour; sitting; workplace; prompts
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prompt group (Experimental): Following an education session on the health benefits of breaking prolonged sitting, the prompt group will receive hourly prompts on their PC to stand. The prompts will be delivered by Microsoft Outlook and will run for a period of 10 weeks. The messages will be short in length, varied and centre around the key message of breaking prolonged sitting by standing.
  Interventions: Behavioral: Hourly prompts to stand delivered by Microsoft Outlook
- Control group (No Intervention): The control group will receive the same education session as the prompt group, but will receive no prompts on their PC.

INTERVENTIONS:
Behavioral: Hourly prompts to stand delivered by Microsoft Outlook
  Arms: Prompt group

SUMMARY:
This study aims to investigate whether hourly prompts, delivered by Microsoft Office onto the PC's of office workers, is effective at reducing unhealthy patterns of sedentary behaviour .

DETAILED DESCRIPTION:
The health benefits of physical activity are widely recognised and there is increasing evidence to show the detrimental effects of sedentary behaviour on health. Both total sedentary time and the temporal pattern of accumulation of sedentary behaviour have a significant effect on health, with prolonged, unbroken periods of sitting being most harmful. Working adults spend a considerable proportion of time in the work domain and there is a high level of prolonged sedentary behaviour in many workplaces .

There is limited evidence from small-scale studies that workplace interventions can reduce prolonged sedentary behaviour of office workers. Providing advice to stand at regular intervals during the working day and using passive computer-based prompts, significantly reduced prolonged sitting by 40 minutes per day and increased self-reported energy expenditure . This indicates that there is potential for resource-light interventions to change behaviour in the workplace, however, evidence for effectiveness, feasibility and acceptability is currently limited.

This proposal is part of an ongoing collaboration with NHS Greater Glasgow & Clyde Healthy Working lives. Representatives from 10 organisations involved with the Healthy Working Lives initiative were previously consulted to find an intervention acceptable to employers and identify companies interested in participating in a pilot study. The consultations generated considerable interest in the project and use of the outlook calendar (available to many staff) to provide prompts to stand-up as an intervention was considered acceptable to many employers. This pilot intervention will therefore build on the group's existing research.

30 desk-based employees will be recruited as participants via an email invitation and the use of posters displayed in the office. Volunteers will be screened regarding inclusion/exclusion criteria given a participant information sheet and asked to provide signed consent.

The study will be a 2-arm RCT of 30 participants split equally between a control and intervention group, where both groups receive education on why and how to reduce prolonged sitting, but the intervention group also receives hourly prompts to stand for a period of 10 weeks. Participants will be randomly assigned to a group either on an individual basis or in clusters by physical location within the office (to minimise the influence of neighbouring colleagues should they be in a different group). The method of randomisation will be decided upon once individuals have volunteered and been screened. Activity monitoring will be made at baseline (before the education session) at week 10 of the intervention and 3 months post-intervention (week 22). All participants will be asked to complete a questionnaire to ascertain basic demographic data, knowledge of and attitudes towards sedentary behaviour and previous engagement with health promotion initiatives. They will then be asked to wear a water-proofed ActivPal monitor on the front of their thigh for a period of 7 days (24 hours a day) in order to measure patterns of sedentary behaviour at baseline. To accompany this measurement they will also keep a diary recording waking and working hours for the same 7 day period.

Following baseline measurements all participants will attend an education session which will cover: what sedentary behaviour is (and how it is different to physical activity), the health problems associated with prolonged sedentary behaviour, how much sitting is recommended and advice on how to reduce and break up prolonged sitting.

Participants will then be randomly assigned (using sealed envelopes prepared by a researcher not involved in recruitment or intervention implementation) to either a control or intervention group so that each group contains 15 participants and, where possible, are physically separated within the office. The control group will return to work as normal following the education session, whereas the intervention group will have a series of prompts uploaded onto their Microsoft Office calendar, via an excel file, reminding them to stand for a period of one minute, every hour during their working day. These prompts will run for a period of 10 weeks. Participants will be able to dismiss prompts as soon as they appear and can choose whether to stand or remain seated. They will also be able to dismiss groups of prompts accumulated during periods away from the computer. The impact on their work is therefore thought to be minimal. The content of the prompts will be brief, varied and contain a positively framed message. During the last week of the 10 week period, both the control group and intervention group will be asked to once again wear an ActivPal monitor and keep a diary for a period of 7 days.

12 weeks after the end of the intervention period, the 7 day ActivPal and diary measurement will be repeated and semi-structured focus groups will be run with participants and organisational representatives with the aim of exploring the feasibility, acceptability, meaningfulness and effectiveness of the intervention. Focus groups will be recorded using a digital voice recorder, topic guides regarding their content are outlined in annex 6 and annex 7.

The validated ActivPal monitors use the acceleration signal from the thigh to categorise data into sitting/lying, standing and walking, but the primary outcome measures will be total time spent sitting at work, and time spent in prolonged sitting events while at work. Electronic copies of this data will be kept for 10 years, alongside electronic and paper copies of the baseline questionnaire and diaries and audio and transcribed accounts of the focus groups, in line with Glasgow Caledonian University's data protection policies. Physical activity data and basic demographic data will also be kept on a password protected database on a secure server. The data held on the database will not be identifiable. The information collected may be used for further analysis by staff and students in the School of Health and Life Sciences at Glasgow Caledonian University at a later date. Access to the database will be controlled by Dr Ben Stansfield, Reader in the School of Health and Life Sciences.

At the end of the study participants will receive an individual report detailing their patterns of sedentary behaviour before, during and after the intervention. They will also have access to the amalgamated report which will be given to the employer summarising the overall findings including the key outcomes of the focus groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 that are currently employed in an office and whose role is primarily desk-based. Must have regular access to Microsoft Outlook on a daily basis

Exclusion Criteria:

* Those with a pre-existing health condition requiring workplace and/or work practice adjustments (unable to stand on a regular basis) or those who currently have a standing workstation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
total time spent sitting at work | 12 weeks
  total time spent sitting at work will be objectively measured using a tri-axial accelerometer

SECONDARY OUTCOMES:
time spent sitting in prolonged sedentary bouts at work | 12 weeks
  total time spent sitting at work in continuous bouts of at least 30 minutes. These will be objectively measured using a tr-axial accelerometer
number of sitting events at work | 12 weeks
  number of sitting events at work are objectively measured using a tr-axial accelerometer
number of prolonged sitting events at work | 12 weeks
  number of sitting events that last at least 30 minutes at work. These are objectively measured using a tr-axial accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Philippa Dall, PhD, Principal Investigator — Senior Research Fellow
Locations (1):
- Glasgow Caledonian University, Glasgow, United Kingdom

REFERENCES:
- [Background] Global Recommendations on Physical Activity for Health. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK305057/ PMID 26180873
- [Background] Healy GN, Matthews CE, Dunstan DW, Winkler EA, Owen N. Sedentary time and cardio-metabolic biomarkers in US adults: NHANES 2003-06. Eur Heart J. 2011 Mar;32(5):590-7. doi: 10.1093/eurheartj/ehq451. Epub 2011 Jan 11. PMID 21224291
- [Background] Ryan, C. G. et. al. (2011) 'Sitting patterns at work: objective measurement of adherence to current recommendations', Ergonomics, 54 (6), pp.531-538.
- [Background] Evans RE, Fawole HO, Sheriff SA, Dall PM, Grant PM, Ryan CG. Point-of-choice prompts to reduce sitting time at work: a randomized trial. Am J Prev Med. 2012 Sep;43(3):293-7. doi: 10.1016/j.amepre.2012.05.010. PMID 22898122
- [Background] Pedersen SJ, Cooley PD, Mainsbridge C. An e-health intervention designed to increase workday energy expenditure by reducing prolonged occupational sitting habits. Work. 2014;49(2):289-95. doi: 10.3233/WOR-131644. PMID 23787256
- [Background] Grant PM, Ryan CG, Tigbe WW, Granat MH. The validation of a novel activity monitor in the measurement of posture and motion during everyday activities. Br J Sports Med. 2006 Dec;40(12):992-7. doi: 10.1136/bjsm.2006.030262. Epub 2006 Sep 15. PMID 16980531
- [Derived] O'Dolan C, Grant M, Lawrence M, Dall P. A randomised feasibility study to investigate the impact of education and the addition of prompts on the sedentary behaviour of office workers. Pilot Feasibility Stud. 2018 Jan 15;4:33. doi: 10.1186/s40814-017-0226-8. eCollection 2018. PMID 29372071